CLINICAL TRIAL: NCT00223743
Title: Novel Therapies for Essential Tremor - Zonisamide Pilot Study
Brief Title: A Safety/Efficacy Trial of Zonisamide for Essential Tremor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Greater Los Angeles Healthcare System (U.S. Federal Agency)
Collaborators: Ralph M. Parsons Foundation (Other)
Responsible Party: Principal Investigator, Adrian Handforth, MD, Assistant Chief, Neurology, VAMC, VA Greater Los Angeles Healthcare System
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0030
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Essential Tremor
Keywords: essential tremor; zonisamide; clinical trial
MeSH Terms: conditions — Essential Tremor | interventions — Zonisamide

ARMS (1):
- Zonisamide (Experimental): Zonisamide administration and tremor assessment to assess efficacy in reducing essential tremor
  Interventions: Drug: Zonisamide

INTERVENTIONS:
Drug: Zonisamide — study drug initially will taken as one 50-mg tablet a day, then the dose increased by one tablet each two weeks, to no more than 3 tablets (150 mg) taken twice a day.

SUMMARY:
The purpose of this pilot study is to obtain information whether the medication zonisamide reduces tremor in persons with essential tremor and is well tolerated.

DETAILED DESCRIPTION:
Essential tremor is common, affecting about four percent of the population above age 40 years. Of these, about half have troublesome tremor that warrants medical therapy, but only half of these find satisfactory treatment. Thus it can be estimated that about one million Americans have not been able to find adequate therapy for their essential tremor. Presently used medications may fail due to lack of efficacy or tolerance. After encountering anecdotal experience of zonisamide's efficacy for essential tremor we decided to conduct a single-site open-treatment rising-dose study with blinded videotape ratings of tremor. Zonisamide is presently on the market in the United States for epilepsy. Its use in other conditions is experimental.

Healthy participants with bilateral hand tremor will initially sign an IRB-approved informed consent form, then have assessments in a Screening Visit to determine that they are healthy (physical and neurological examinations, routine blood tests, electrocardiogram) and tremor assessments with rating scales. Tremor at each visit will be videotaped, as well as assessed openly by a rater. If participants meet eligibility criteria, they will return to a Baseline Visit (Visit 1) for repeat tremor assessment and the initial dispensation of zonisamide.

The study drug initially will taken as one 50-mg tablet a day, then the dose increased by one tablet each two weeks, to no more than 3 tablets (150 mg) taken twice a day. During this 12-week dose adjustment phase, the participant will be seen in clinic each 4 weeks for tremor assessments and review of health status. In addition, the participant will be contacted by telephone each week. If any symptom occurs suggestive of side effects, the escalation will be stopped or the dose reduced in order to resolve the symptom.

At the end of the 12-week dose adjustment phase, at Visit 4, it will be determined whether meaningful tremor reduction has occurred at the target dose of 300 mg per day or at a lesser but tolerated dose. If not, the participant will discontinue from the study. If benefit has occurred, the subject will be invited to continue taking zonisamide for another 12 weeks, at the conclusion of which the participant will be seen in the final visit (Visit 5).

The videotapes will be coded so that the order they were made is not apparent, and the degree of tremor will be rated by a rater who does not know the study participants.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* diagnosis of essential tremor
* tremor present in both hands for at least one year
* tremor is bothersome in at least one hand, so that reduction of tremor would improve quality of life
* able to comply with study visits and procedures
* has voluntarily signed consent form
* able to abstain from alcohol for 12 hours prior to each visit, and from caffeine on day prior to visit
* taking no medications or stable doses of anti-tremor medication for 4 weeks prior to the Baseline visit

Exclusion Criteria:

* medical condition likely to cause hospitalization during the study
* progressive neurological disorder other than essential tremor
* history of serious psychiatric illness
* history of drug or alcohol abuse in past year
* consumes more than two glasses of wine or equivalent per day
* has received botulinum toxin injection in past 6 months
* currently using experimental device
* has taken experimental drug within 5 half lives of its elimination
* has received deep brain stimulation in past two weeks or has potential need for this therapy during the study
* thalamotomy within the past 6 months
* taking medications judged by investigator to exacerbate tremor
* has probable cause of tremor other than essential tremor
* condition likely to interfere with absorption, metabolism or elimination of study drug
* hepatic disease
* renal disease
* history of renal stones
* history of allergy to sulfonamides

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2004-11; Primary Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
The degree of tremor at the end of the dose adjustment phase compared to baseline. | 3 months

SECONDARY OUTCOMES:
Quality of life. | 6 months
Degree of tremor at the end of the extension phase compared to the beginning of the extension phase. | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Handforth, M.D., Principal Investigator — Veterans Affairs Greater Los Angeles
Locations (1):
- VA Greater Los Angeles, Los Angeles, California, United States